CLINICAL TRIAL: NCT02680496
Title: Energy Consumption and Cardiorespiratory Load During Walking With and Without Robot-Assistance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties patient recruitment
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Nina Lefeber, PhD student, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LOKOMAT STUDY I; SBO-IWT MIRAD project (Other Grant/Funding Number: IWT (120057)); SBO doctoral grant (Other Grant/Funding Number: Research Foundation - Flanders)
Record Dates: First submitted 2016-01-27; First posted 2016-02-11 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Stroke
Keywords: Robot-Assistance; Gait [MeSH]; Energy Consumption; Cardiorespiratory Load; Stroke [MeSH]
MeSH Terms: conditions — Stroke | interventions — Exercise Test

ARMS (6):
- Lokomat - Treadmill - Overground (Experimental): Walking order: lokomat walking, treadmill walking, overground walking
  Interventions: Device: Lokomat; Other: Treadmill; Other: Overground
- Lokomat - Overground - Treadmill (Experimental): Walking order: lokomat walking, overground walking, treadmill walking
  Interventions: Device: Lokomat; Other: Treadmill; Other: Overground
- Treadmill - Lokomat - Overground (Experimental): Walking order: treadmill walking, lokomat walking, overground walking
  Interventions: Device: Lokomat; Other: Treadmill; Other: Overground
- Treadmill - Overground - Lokomat (Experimental): Walking order: treadmill walking, overground walking, lokomat walking
  Interventions: Device: Lokomat; Other: Treadmill; Other: Overground
- Overground - Lokomat - Treadmill (Experimental): Walking order: overground walking, lokomat walking, treadmill walking
  Interventions: Device: Lokomat; Other: Treadmill; Other: Overground
- Overground - Treadmill - Lokomat (Experimental): Walking order: overground walking, treadmill walking, lokomat walking
  Interventions: Device: Lokomat; Other: Treadmill; Other: Overground

INTERVENTIONS:
Device: Lokomat — A single walking trial in which the patient walks in the Lokomat with 60% guidance force for 30 minutes at comfortable walking speed (body-weight supported if necessary)
Other: Treadmill — A single walking trial in which the patient walks on a treadmill for 30 minutes at comfortable walking speed (body-weight supported if necessary)
Other: Overground — A single walking trial in which the patient walks overground for 30 minutes at comfortable walking speed (body-weight supported if necessary)

SUMMARY:
The primary objective of the study is to investigate the energy consumption, cardiorespiratory load and perceived exertion, and how these parameters change, during walking with robot-assistance compared to walking on a treadmill and walking overground in stroke patients.

A secondary objective is to investigate whether these changes or differences in energy consumption, cardiorespiratory load and perceived exertion during walking with and without robot-assistance in stroke patients are related to changes or differences spatiotemporal gait characteristics.

DETAILED DESCRIPTION:
Background. Impaired cardiorespiratory fitness, which is a major risk factor in the development of cardiorespiratory diseases, is frequently reported in stroke patients. The mean energy cost of walking, i.e. the amount of oxygen consumption in milliliter per kilogram of body-weight per meter, in stroke patients is almost twice as high compared to healthy subjects (resp. 0.27 ml/kg/m vs. 0.15 ml/kg/m). In the rehabilitation of stroke patients, the primary aim is to improve kinematic and functional gait-related parameters. However, due to the previously mentioned cardiorespiratory risks, it is important to be aware of the energy consumption and cardiorespiratory load of stroke patients during gait rehabilitation. In the past, gait training was mainly fulfilled by treadmill training, overground training and/or more conventional therapies, but in recent years, the implementation of robot-assistance in gait rehabilitation is increasing. However, what the influence is of robot-assistance on the cardiorespiratory load and energy consumption, and therefore also what potentially negative and/or positive side effects are for the cardiorespiratory system, is less investigated and unclear.

Up to now, short walking durations of robot-assisted gait (up to 7 minutes) seem less energy consuming and cardiorespiratory stressful than walking without robot-assistance. However, what the influences are of longer walking durations is not clear. In addition, it is also unclear why possible differences between robot-assisted gait and walking without robot-assistance might exist. One possible explanation might be that differences in spatiotemporal gait parameters are responsible for differences in energy consumption and cardiorespiratory load.

Patient recruitment. Stroke patients in the Rehabilitation Centre St. Ursula (Herk-de-Stad, Belgium) will receive verbal and written information on the aims and interventions of the study. Eligible stroke patients, who agree to participate in the study, will be recruited. Signed informed consent will be obtained from all participants.

Sample size. Sample size calculation is based on previous investigations indicating large effect sizes between the effect of robot-assisted gait compared to walking without robot-assistance on energy consumption and cardiorespiratory load (based on a systematic review submitted for peer-review). To detect a large effect size (f = 0.40) of robot-assisted gait compared to overground and treadmill gait on energy consumption, cardiorespiratory load and perceived fatigue, in a repeated measures within subjects design (3 walking conditions and 4 measurements), with a significance level of 5% and a power level of 80%, a sample size of 21 subjects is needed (G*Power 3.1 for Mac). Sample size is inflated up to 24 subjects, so each walking order will be performed the same number of times.

Intervention. Patients will be tested in 3 single walking sessions each on a separate day: walking in the Lokomat with 60% guidance force, walking on a treadmill and walking overground. Within subjects, all walking conditions will be performed at the same comfortable walking speed (CWS), with the same amount of body-weight support (BWS) (if necessary) during a total duration of maximum 30 minutes. The CWS (with a maximum of 3.2 kmph corresponding to the maximum Lokomat speed) and the amount of BWS (if necessary) will be individually determined on a separate day before the start of the study. Walking tests will be terminated early when relative or absolute indications are presented as reported by the American Heart Association or when patients are unable to continue walking. Patients will be asked to not consume food, alcohol, caffeine or nicotine at least 3 hours prior to the intervention, and not to perform additional strenuous activities at least 12 hours prior to the interventions. Walking sessions will be controlled for time of day. Before the start of the study, demographic and clinical characteristics will be collected and the CWS and the amount of BWS (if necessary) will be determined in a 10 minute walking test. At the start of each walking condition, a chest-carrying gas analysis system with mouth mask (Metamax 3B, Cortex, Germany), a heart rate belt (Polar H7) and 2 wearable foot sensors (Physiolog, Gait Up, Switzerland) will be applied. Patients will be seated for 5 minutes during which resting values (energy consumption, cardiorespiratory parameters and perceived fatigue) will be registered. After a resting period of 5 minutes, patients will walk for 30 minutes during which energy consumption, cardiorespiratory parameters, perceived fatigue and spatiotemporal parameters will be monitored continuously. Perceived fatigue will be registered every minute. Average values at rest, the beginning, middle and end of the walking sessions will be calculated offline.

Randomization and Concealment. Walking sessions will be performed in a random order at 3 separate days. An independent investigator will assign the 24 patients (in 2 series of 12) at random to one of the 6 possible walking orders using a random sequence generator. Allocation will be concealed for the investigators using an excel file with blind and locked sections, to which only the independent investigator has access to. The random walking order of the patient will therefore only be available when the patient has been recruited and his name is entered in the excel sheet. This method will assure that the investigator does not know the walking order of the next participant.

Dropout. In case subjects drop out, the subject will be replaced by a new participant who will perform all three trials in the same randomized order as the subject that dropped out. So, in case of drop out, additional patients will be tested until the data of 24 patients that participated in all three conditions are collected.

Statistical analysis. Statistics will be performed using SPSS (IBM, Chicago, IL). Descriptive statistics will be calculated for baseline demographic and clinical patient characteristics. Repeated measures analyses of variance (ANOVA) with Bonferroni correction for multiple comparisons will be used to analyze differences in primary and secondary outcomes within and between walking conditions. Regression analysis will be performed to evaluate whether (changes in) spatiotemporal parameters are predictive for (changes in) energy consumption. The significance level will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients with a lower limb motor impairment
* Time since stroke < 1 year
* ≥ 18 years
* < 193 cm
* < 135kg
* Able to walk overground (body-weight support allowed if necessary) for at least 10 minutes at a comfortable walking speed

Exclusion Criteria:

* Contra-indications for exercise testing according to the American College of Sports Medicine
* Musculoskeletal problems (other than stroke) affecting the ability to walk
* Concurrent pulmonary diseases
* Concurrent neurological diseases
* Communicative and/or cognitive problems affecting the ability to comprehend or follow instructions
* Other problems that affect the execution of the interventions, e.g. severe spasticity, contractures or dermatologic contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Gross oxygen consumption (VO2) at rest | Minute 5 of 5-minute resting period
  Average oxygen consumption (mL/kg/min). Oxygen consumption will be measured continuously (from the beginning of rest till the end of walking). Offline calculations (e.g. averages) will be performed afterwards.
Gross oxygen consumption (VO2) at begin of walking | Minute 6 of 30-minute walking period
  Average oxygen consumption (mL/kg/min). Oxygen consumption will be measured continuously (from the beginning of rest till the end of walking). Offline calculations (e.g. averages) will be performed afterwards.
Gross oxygen consumption (VO2) at mid of walking | Minute 18 of 30-minute walking period
  Average oxygen consumption (mL/kg/min). Oxygen consumption will be measured continuously (from the beginning of rest till the end of walking). Offline calculations (e.g. averages) will be performed afterwards.
Gross oxygen consumption (VO2) at end of walking | Minute 30 of 30-minute walking period
  Average oxygen consumption (mL/kg/min). Oxygen consumption will be measured continuously (from the beginning of rest till the end of walking). Offline calculations (e.g. averages) will be performed afterwards.
Net oxygen consumption (VO2) | Change between average VO2 at minute 5 of rest and minute 6 of walking, at minute 5 of rest and minute 18 of walking, at minute 5 of rest and minute 30 of walking
  Change in average oxygen consumption (mL/kg/min) at different time frames during walking compared to rest. VO2 will be measured continuously (from the beginning of rest till the end of walking). Offline calculations will be performed afterwards.
Gross minute ventilation (VE) at rest | Minute 5 of 5-minute resting period
  Average amount of air in- or exhaled (L/min). VE will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross minute ventilation (VE) at begin of walking | Minute 6 of 30-minute walking period
  Average amount of air in- or exhaled (L/min). VE will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross minute ventilation (VE) at mid of walking | Minute 18 of 30-minute walking period
  Average amount of air in- or exhaled (L/min). VE will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross minute ventilation (VE) at end of walking | Minute 30 of 30-minute walking period
  Average amount of air in- or exhaled (L/min). VE will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Net minute ventilation (VE) | Change between average VE at minute 5 of rest and minute 6 of walking, at minute 5 of rest and minute 18 of walking, at minute 5 of rest and minute 30 of walking
  Change in average amount of air in- or exhaled (L/min) at different time frames during walking compared to rest. VE will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross respiration rate (RR) at rest | Minute 5 of 5-minute resting period
  Average breaths per minute. Respiration rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross respiration rate (RR) at begin of walking | Minute 6 of 30-minute walking period
  Average breaths per minute. Respiration rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross respiration rate (RR) at mid of walking | Minute 18 of 30-minute walking period
  Average breaths per minute. Respiration rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross respiration rate (RR) at end of walking | Minute 30 of 30-minute walking period
  Average breaths per minute. Respiration rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Net respiration rate (RR) | Change between average respiration rate at minute 5 of rest and minute 6 of walking, at minute 5 of rest and minute 18 of walking, at minute 5 of rest and minute 30 of walking
  Change in respiration rate (breaths per minute) at different time frames during walking compared to rest. Respiration rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross heart rate (HR) at rest | Minute 5 of 5-minute resting period
  Average heart rate (beats/min). Heart rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross heart rate (HR) at begin of walking | Minute 6 of 30-minute walking period
  Average heart rate (beats/min). Heart rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross heart rate (HR) at mid of walking | Minute 18 of 30-minute walking period
  Average heart rate (beats/min). Heart rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross heart rate (HR) at end of walking | Minute 30 of 30-minute walking period
  Average heart rate (beats/min). Heart rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Net heart rate (HR) | Change between average heart rate at minute 5 of rest and minute 6 of walking, at minute 5 of rest and minute 18 of walking, at minute 5 of rest and minute 30 of walking
  Change in average heart rate (beats/min) at different time frames during walking compared to rest. Heart rate will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Gross Respiratory Exchange Ratio (RER) at rest | Minute 5 of 5-minute resting period
  RER is the ratio between the amount of CO2 produced by the body and the amount of VO2 consumed by the body (VCO2/VO2). This ratio gives an indication of the type of fuel used to produce ATP.
Gross Respiratory Exchange Ratio (RER) at begin of walking | Minute 6 of 30-minute walking period
  RER is the ratio between the amount of CO2 produced by the body and the amount of VO2 consumed by the body (VCO2/VO2). This ratio gives an indication of the type of fuel used to produce ATP.
Gross Respiratory Exchange Ratio (RER) at mid of walking | Minute 18 of 30-minute walking period
  RER is the ratio between the amount of CO2 produced by the body and the amount of VO2 consumed by the body (VCO2/VO2). This ratio gives an indication of the type of fuel used to produce ATP.
Gross Respiratory Exchange Ratio (RER) at end of walking | Minute 30 of 30-minute walking period
  RER is the ratio between the amount of CO2 produced by the body and the amount of VO2 consumed by the body (VCO2/VO2). This ratio gives an indication of the type of fuel used to produce ATP.
Net Respiratory Exchange Ratio (RER) | Change between average RER at minute 5 of rest and minute 6 of walking, at minute 5 of rest and minute 18 of walking, at minute 5 of rest and minute 30 of walking
  Change in RER at different time frames during walking compared to rest. RER will be measured continuously (from the beginning of rest till the end of the walking session). Offline calculations will be performed afterwards.
Metabolic Equivalent of Task (MET) at begin of walking | Minute 6 of 30-minute walking period
  Expression of the intensity of physical activity (at different time frames) defined as oxygen consumption during walking divided by reference oxygen consumption in rest. Oxygen consumption will be measured continuously (from the beginning of rest till the end of walking). Offline calculations will be performed afterwards.
Metabolic Equivalent of Task (MET) at mid of walking | Minute 18 of 30-minute walking period
  Expression of the intensity of physical activity (at different time frames) defined as oxygen consumption during walking divided by reference oxygen consumption in rest. Oxygen consumption will be measured continuously (from the beginning of rest till the end of walking). Offline calculations will be performed afterwards.
Metabolic Equivalent of Task (MET) at end of walking | Minute 30 of 30-minute walking period
  Expression of the intensity of physical activity (at different time frames) defined as oxygen consumption during walking divided by reference oxygen consumption in rest. Oxygen consumption will be measured continuously (from the beginning of rest till the end of walking). Offline calculations will be performed afterwards

SECONDARY OUTCOMES:
Gross perceived exertion (assessed by the 6-20 Borg scale) at rest | Minute 5 of 5-minute resting period
  Rating of perceived effort, strain and/or fatigue pointed on a 15-point Borg scale (6-20). Borg score will be measured at the end of rest (min 5) and at the end of every minute of walking.
Gross perceived exertion (assessed by the 6-20 Borg scale) at begin of walking | Minute 6 of 30-minute walking period
  Rating of perceived effort, strain and/or fatigue pointed on a 15-point Borg scale (6-20). Borg score will be measured at the end of rest (min 5) and at the end of every minute of walking.
Gross perceived exertion (assessed by the 6-20 Borg scale) at mid of walking | Minute 18 of 30-minute walking period
  Rating of perceived effort, strain and/or fatigue pointed on a 15-point Borg scale (6-20). Borg score will be measured at the end of rest (min 5) and at the end of every minute of walking.
Gross perceived exertion (assessed by the 6-20 Borg scale) at end of walking | Minute 30 of 30-minute walking period
  Rating of perceived effort, strain and/or fatigue pointed on a 15-point Borg scale (6-20). Borg score will be measured at the end of rest (min 5) and at the end of every minute of walking.
Net perceived exertion (assessed by the 6-20 Borg scale) | Change between Borg score at minute 5 of rest and minute 6 of walking, at minute 5 of rest and minute 18 of walking, at minute 5 of rest and minute 30 of walking
  Change in Borg score at different time frames during walking compared to rest. Borg score will be measured at the end of rest (min 5) and at the end of every minute of walking.
Total walking duration | Begin till end of walking (up to 30 minutes)
  Total walking duration the patient can achieve in a single walking session (with a maximum of 30 minutes)

OTHER OUTCOMES:
Paretic cadence | Minute 6, 18 and 30 of 30-minute walking period
  The average amount of steps per minute at the paretic side at different time frames. Cadence will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic cadence | Minute 6, 18 and 30 of 30-minute walking period
  The average amount of steps per minute at the paretic side at different time frames. Cadence will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Cadence symmetry ratio | Minute 6, 18 and 30 of 30-minute walking period
  The ratio of paretic and non-paretic cadence with the numerator always being the greater of the two values, so that results are not skewed by values <1.0 (1.0 indicating perfect symmetry). Direction of asymmetry will be retained with a sign convention (e.g. +/- to indicate favoring of the paretic/non-paretic limb, respectively).
Paretic cadence variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in paretic cadence between consecutive gait cycles. Cadence will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic cadence variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in non-paretic cadence between consecutive gait cycles. Cadence will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Paretic gait cycle time | Minute 6, 18 and 30 of 30-minute walking period
  The average duration of a gait cycle (expressed in seconds) at the paretic side at different time frames. Gait cycle time will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic gait cycle time | Minute 6, 18 and 30 of 30-minute walking period
  The average duration of a gait cycle (expressed in seconds) at the non-paretic side at different time frames. Gait cycle time will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Gait cycle time asymmetry ratio | Minute 6, 18 and 30 of 30-minute walking period
  The ratio of paretic and non-paretic gait cycle time with the numerator always being the greater of the two values, so that results are not skewed by values <1.0 (1.0 indicating perfect symmetry). Direction of asymmetry will be retained with a sign convention (e.g. +/- to indicate favoring of the paretic/non-paretic limb, respectively).
Paretic gait cycle time variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in paretic gait cycle time between consecutive gait cycles. Gait cycle time will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic gait cycle time variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in non-paretic gait cycle time between consecutive gait cycles. Gait cycle time will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Paretic stance | Minute 6, 18 and 30 of 30-minute walking period
  The average portion of the cycle during which part of the paretic foot touches the ground (expressed in % of cycle duration) at different time frames. Stance ratio will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic stance | Minute 6, 18 and 30 of 30-minute walking period
  The average portion of the cycle during which part of the non-paretic foot touches the ground (expressed in % of cycle duration) at different time frames. Stance ratio will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Stance symmetry ratio | Minute 6, 18 and 30 of 30-minute walking period
  The ratio of paretic and non-paretic stance with the numerator always being the greater of the two values, so that results are not skewed by values <1.0 (1.0 indicating perfect symmetry). Direction of asymmetry will be retained with a sign convention (e.g. +/- to indicate favoring of the paretic/non-paretic limb, respectively).
Paretic stance variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in paretic stance between consecutive gait cycles. Stance will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic stance variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in non-paretic stance between consecutive gait cycles. Stance will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Paretic swing | Minute 6, 18 and 30 of 30-minute walking period
  The average portion of the gait cycle during which the paretic foot is in the air and does not touch the ground (expressed in % of gait cycle) at different time frames. Swing ratio will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic swing | Minute 6, 18 and 30 of 30-minute walking period
  The average portion of the gait cycle during which the non-paretic foot is in the air and does not touch the ground (expressed in % of gait cycle) at different time frames. Swing ratio will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Swing symmetry ratio | Minute 6, 18 and 30 of 30-minute walking period
  The ratio of paretic and non-paretic swing with the numerator always being the greater of the two values, so that results are not skewed by values <1.0 (1.0 indicating perfect symmetry). Direction of asymmetry will be retained with a sign convention (e.g. +/- to indicate favoring of the paretic/non-paretic limb, respectively).
Paretic swing variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in paretic swing between consecutive gait cycles. Swing will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic swing variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in non-paretic swing between consecutive gait cycles. Swing will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Double support | Minute 6, 18 and 30 of 30-minute walking period
  The average portion of the cycle during which both feet touch the ground (expressed in % of cycle duration) at different time frames. Double support will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Double support variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in double support between consecutive gait cycles. Double support will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Paretic stride length | Minute 6, 18 and 30 of 30-minute walking period
  The average distance (expressed in meters) between two successive paretic footprints on the ground, from the heel of the paretic foot to the heel of the paretic foot, one cycle after, at different time frames. Stride length will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic stride length | Minute 6, 18 and 30 of 30-minute walking period
  The average distance (expressed in meters) between two successive non-paretic footprints on the ground, from the heel of the non-paretic foot to the heel of the non-paretic foot, one cycle after, at different time frames. Stride length will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Stride length symmetry ratio | Minute 6, 18 and 30 of 30-minute walking period
  The ratio of paretic and non-paretic stride length with the numerator always being the greater of the two values, so that results are not skewed by values <1.0 (1.0 indicating perfect symmetry). Direction of asymmetry will be retained with a sign convention (e.g. +/- to indicate favoring of the paretic/non-paretic limb, respectively).
Paretic stride length variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in paretic stride length between consecutive gait cycles. Stride length will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.
Non-paretic stride length variability | Minute 6, 18 and 30 of 30-minute walking period
  The average intra-subject variation in non-paretic stride length between consecutive gait cycles. Stride length will be measured continuously (from the beginning till the end of walking). Offline calculations will be performed afterwards.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kerckhofs, Prof. PhD, Study Chair — Vrije Universiteit Brussel; Eva Swinnen, PhD, Study Director — Vrije Universiteit Brussel; Nina Lefeber, PhD student, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- St. Ursula Rehabilitation Centre (Jessa Hospital), Herk-de-Stad, Limburg, Belgium

REFERENCES:
- [Background] Myers J, McAuley P, Lavie CJ, Despres JP, Arena R, Kokkinos P. Physical activity and cardiorespiratory fitness as major markers of cardiovascular risk: their independent and interwoven importance to health status. Prog Cardiovasc Dis. 2015 Jan-Feb;57(4):306-14. doi: 10.1016/j.pcad.2014.09.011. Epub 2014 Sep 28. PMID 25269064
- [Background] Kelly JO, Kilbreath SL, Davis GM, Zeman B, Raymond J. Cardiorespiratory fitness and walking ability in subacute stroke patients. Arch Phys Med Rehabil. 2003 Dec;84(12):1780-5. doi: 10.1016/s0003-9993(03)00376-9. PMID 14669183
- [Background] Smith AC, Saunders DH, Mead G. Cardiorespiratory fitness after stroke: a systematic review. Int J Stroke. 2012 Aug;7(6):499-510. doi: 10.1111/j.1747-4949.2012.00791.x. Epub 2012 May 9. PMID 22568786
- [Background] Waters RL, Mulroy S. The energy expenditure of normal and pathologic gait. Gait Posture. 1999 Jul;9(3):207-31. doi: 10.1016/s0966-6362(99)00009-0. PMID 10575082
- [Background] Mehrholz J, Pohl M, Elsner B. Treadmill training and body weight support for walking after stroke. Cochrane Database Syst Rev. 2014 Jan 23;2014(1):CD002840. doi: 10.1002/14651858.CD002840.pub3. PMID 24458944
- [Background] States RA, Salem Y, Pappas E. Overground gait training for individuals with chronic stroke: a Cochrane systematic review. J Neurol Phys Ther. 2009 Dec;33(4):179-86. doi: 10.1097/NPT.0b013e3181c29a8c. PMID 20208461
- [Background] Swinnen E, Duerinck S, Baeyens JP, Meeusen R, Kerckhofs E. Effectiveness of robot-assisted gait training in persons with spinal cord injury: a systematic review. J Rehabil Med. 2010 Jun;42(6):520-6. doi: 10.2340/16501977-0538. PMID 20549155
- [Background] Swinnen E, Beckwee D, Pinte D, Meeusen R, Baeyens JP, Kerckhofs E. Treadmill training in multiple sclerosis: can body weight support or robot assistance provide added value? A systematic review. Mult Scler Int. 2012;2012:240274. doi: 10.1155/2012/240274. Epub 2012 May 30. PMID 22701177
- [Background] Mehrholz J, Elsner B, Werner C, Kugler J, Pohl M. Electromechanical-assisted training for walking after stroke. Cochrane Database Syst Rev. 2013 Jul 25;2013(7):CD006185. doi: 10.1002/14651858.CD006185.pub3. PMID 23888479
- [Background] Ada L, Dean CM, Vargas J, Ennis S. Mechanically assisted walking with body weight support results in more independent walking than assisted overground walking in non-ambulatory patients early after stroke: a systematic review. J Physiother. 2010;56(3):153-61. doi: 10.1016/s1836-9553(10)70020-5. PMID 20795921
- [Background] David D, Regnaux JP, Lejaille M, Louis A, Bussel B, Lofaso F. Oxygen consumption during machine-assisted and unassisted walking: a pilot study in hemiplegic and healthy humans. Arch Phys Med Rehabil. 2006 Apr;87(4):482-9. doi: 10.1016/j.apmr.2005.11.034. PMID 16571386
- [Background] Delussu AS, Morone G, Iosa M, Bragoni M, Traballesi M, Paolucci S. Physiological responses and energy cost of walking on the Gait Trainer with and without body weight support in subacute stroke patients. J Neuroeng Rehabil. 2014 Apr 10;11:54. doi: 10.1186/1743-0003-11-54. PMID 24720844
- [Background] Farris RJ, Quintero HA, Murray SA, Ha KH, Hartigan C, Goldfarb M. A preliminary assessment of legged mobility provided by a lower limb exoskeleton for persons with paraplegia. IEEE Trans Neural Syst Rehabil Eng. 2014 May;22(3):482-90. doi: 10.1109/TNSRE.2013.2268320. Epub 2013 Jun 18. PMID 23797285
- [Background] Fenuta AM, Hicks AL. Metabolic demand and muscle activation during different forms of bodyweight supported locomotion in men with incomplete SCI. Biomed Res Int. 2014;2014:632765. doi: 10.1155/2014/632765. Epub 2014 May 21. PMID 24971340
- [Background] Kitatani R, Ohata K, Takahashi H, Shibuta S, Hashiguchi Y, Yamakami N. Reduction in energy expenditure during walking using an automated stride assistance device in healthy young adults. Arch Phys Med Rehabil. 2014 Nov;95(11):2128-33. doi: 10.1016/j.apmr.2014.07.008. Epub 2014 Jul 24. PMID 25064779
- [Background] Maeshima S, Osawa A, Nishio D, Hirano Y, Takeda K, Kigawa H, Sankai Y. Efficacy of a hybrid assistive limb in post-stroke hemiplegic patients: a preliminary report. BMC Neurol. 2011 Sep 27;11:116. doi: 10.1186/1471-2377-11-116. PMID 21943320
- [Background] Malcolm P, Derave W, Galle S, De Clercq D. A simple exoskeleton that assists plantarflexion can reduce the metabolic cost of human walking. PLoS One. 2013;8(2):e56137. doi: 10.1371/journal.pone.0056137. Epub 2013 Feb 13. PMID 23418524
- [Background] van Nunen MP, Gerrits KH, de Haan A, Janssen TW. Exercise intensity of robot-assisted walking versus overground walking in nonambulatory stroke patients. J Rehabil Res Dev. 2012;49(10):1537-46. doi: 10.1682/jrrd.2011.12.0252. PMID 23516057
- [Background] Israel JF, Campbell DD, Kahn JH, Hornby TG. Metabolic costs and muscle activity patterns during robotic- and therapist-assisted treadmill walking in individuals with incomplete spinal cord injury. Phys Ther. 2006 Nov;86(11):1466-78. doi: 10.2522/ptj.20050266. PMID 17079746
- [Background] Hornby TG, Kinnaird CR, Holleran CL, Rafferty MR, Rodriguez KS, Cain JB. Kinematic, muscular, and metabolic responses during exoskeletal-, elliptical-, or therapist-assisted stepping in people with incomplete spinal cord injury. Phys Ther. 2012 Oct;92(10):1278-91. doi: 10.2522/ptj.20110310. Epub 2012 Jun 14. PMID 22700537
- [Background] Krewer C, Muller F, Husemann B, Heller S, Quintern J, Koenig E. The influence of different Lokomat walking conditions on the energy expenditure of hemiparetic patients and healthy subjects. Gait Posture. 2007 Sep;26(3):372-7. doi: 10.1016/j.gaitpost.2006.10.003. Epub 2006 Nov 20. PMID 17113774
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] Patterson KK, Gage WH, Brooks D, Black SE, McIlroy WE. Evaluation of gait symmetry after stroke: a comparison of current methods and recommendations for standardization. Gait Posture. 2010 Feb;31(2):241-6. doi: 10.1016/j.gaitpost.2009.10.014. Epub 2009 Nov 22. PMID 19932621